CLINICAL TRIAL: NCT01856530
Title: Effect of Oxytocin on Pro-Social Behavior in Social Anxiety Disorder
Brief Title: Effect of Oxytocin Nasal Sprays on Social Behavior in Social Anxiety Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stefan G. Hofmann (Other)
Responsible Party: Sponsor-Investigator, Stefan G. Hofmann, Principal Investigator, Boston University Charles River Campus
Organization: Boston University Charles River Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-31668
Record Dates: First submitted 2013-05-10; First posted 2013-05-17 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): Liquid intranasal oxytocin, 24 IU, administered once
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Matched placebo nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Liquid metered-dose nasal spray, 24 IU, administered once
  Arms: Oxytocin
Drug: Placebo — Matched placebo nasal spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn more about how the hormone, oxytocin, impacts social behavior in terms of cooperation with others, attention processing, and reward processing, among patients with social anxiety disorder. Based on available research, the investigators predict that in patients with social anxiety disorder, oxytocin will improve social cooperation during an online ball-tossing game called Cyberball, reduce attention toward socially threatening cues during a dot-probe task, and lead to greater willingness to work for monetary rewards for others rather than themselves during an effort expenditure task.

ELIGIBILITY:
Inclusion Criteria:

* Males > 18 years of age with a primary (or co-principal) psychiatric diagnosis of social anxiety disorder (SAD), as defined by Diagnostic and Statistical Manual-IV (DSM-IV) criteria;
* Current Liebowitz Social Anxiety Scale (LSAS) score > 60, which is a clinical threshold for SAD symptoms;
* Comorbid present DSM-IV Major Depression, Dysthymia, Specific Phobia, or any of the other anxiety disorders as diagnosed by DSM-IV criteria will be permitted as long as SAD is primary (the disorder that is most distressing to the patient). Inclusion of patients with comorbidity will permit accrual of a more clinically relevant patient population;
* Willingness to participate in and comply with the study procedures as indicated by signing the informed consent form.

Exclusion Criteria:

* Subjects with a serious medical illness for which hospitalization may be likely within the next three months;
* Subjects with a current diagnosis of schizophrenia, psychotic disorders, bipolar disorder, mental disorder due to a medical condition or substance, substance abuse or dependence, as diagnosed by DSM-IV criteria;
* Concurrent use of other psychotropic medications is excluded, except for antidepressants that have been taken at a stable dose for at least 2 weeks;
* Active suicidal or homicidal ideation or suicide attempts within the past six months requiring hospitalization;
* Subjects with significant nasal pathology (atrophic rhinitis, recurrent nose bleeds, or history of hypophysectomy);
* Smokers who smoke more than 15 cigarettes per day;
* Those who smoke cigarettes or have caffeine or alcohol within 24 hours of the study visit.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Anxiety and Related Disorders at Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fang A, Treadway MT, Hofmann SG. Working hard for oneself or others: Effects of oxytocin on reward motivation in social anxiety disorder. Biol Psychol. 2017 Jul;127:157-162. doi: 10.1016/j.biopsycho.2017.05.015. Epub 2017 May 27. PMID 28559206

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 60 participants were enrolled in the study, 6 participants were found to be ineligible due to meeting criteria for substance dependence (n=2), a primary diagnosis of posttraumatic stress disorder (n=1), and not meeting criteria for social anxiety disorder (n=3). Therefore, only 54 participants were assigned to groups.
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 27 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 19 | 16 | 35
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Social Cooperation
Description: The outcome measure involved difference scores in the number of balls tossed to Player 1 between two conditions of the task. Across both conditions, the participant (always assigned as "Player 2") played with 3 other on-line players in real time. In Condition 1, Player 1 was programmed to toss on average 70% of his balls to the participant. In Condition 2, Player 1's behavior switched such that he was programmed to toss on average only 10% of his balls to the participant. The data reported below is the number of balls tossed to Player 1 in Condition 2 minus balls tossed under Condition 1.
Time Frame: Day 1 (first day oxytocin or placebo was administered)
Population: Data from 2 participants could not be analyzed due to technical difficulties with the computer task. Thus, the number of participants analyzed was 52 in total, rather than 54.
Measure: Mean (Standard Deviation); unit: Ball tosses
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 26 | 26
Ball tosses | 4.42 (6.706) | 4.69 (6.078)

2. Primary Outcome: Disengagement From Social Threat Cues
Description: The outcome measure involved difference scores in response latencies on disengagement trials for disgust versus neutral cues. Difference scores were calculated as response latencies during disengagement trials for disgust cues minus response latencies during disengagement trials for neutral cues. Negative change scores represent an improvement in disengagement.
Time Frame: Day 1 (first day oxytocin or placebo was administered)
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 27 | 27
Milliseconds | 1.34 (36.79) | -2.69 (52.39)

3. Secondary Outcome: Perceived Trust Scores on a 1-7 Likert Scale
Description: Participants will rate their perceived level of trust (on a 1-7 Likert scale) toward Player 1 during online ball-tossing task. Higher ratings on this scale reflect greater perceived trust toward Player 1.
Time Frame: Day 1 (first day oxytocin or placebo was administered)
Population: Due to technical difficulties during the computer task, two participants did not complete this questionnaire and were not included in the analysis. Thus, only 52 participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 26 | 26
units on a scale | 4.65 (1.47) | 4.73 (1.12)

4. Secondary Outcome: Perceived Empathy Scores on a 1-7 Likert Scale
Description: Participants will rate their level of perceived empathy (on a 1-7 Likert scale) with Player 1 during online ball-tossing task. Higher scores on this scale reflect greater perceived empathy toward Player 1.
Time Frame: Day 1 (first day oxytocin or placebo was administered)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 26 | 26
units on a scale | 4.46 (1.39) | 4.27 (1.46)

5. Secondary Outcome: Perceived Preference Scores on a 1-7 Likert Scale
Description: Participants will rate their level of preference (on a 1-7 Likert scale) for Player 1 during online ball-tossing task. Higher scores on this scale reflect greater preference for Player 1.
Time Frame: Day 1 (first day oxytocin or placebo was administered)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 26 | 26
units on a scale | 5.04 (1.40) | 5.04 (1.18)

6. Secondary Outcome: Perceived Rejection Scores on a 1-7 Likert Scale
Description: Participants will rate their level of perceived rejection (on a 1-7 Likert scale) from Player 1 during online ball-tossing task. Higher scores on this scale reflect greater perceived rejection from Player 1.
Time Frame: Day 1 (first day oxytocin or placebo was administered)
Population: Due to technical difficulties during the computer task, two participants did not complete this questionnaire and were not included in this analysis. Thus, only 52 participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 26 | 26
units on a scale | 3.35 (1.41) | 3.65 (1.29)

ADVERSE EVENTS:
Arm/Group | Oxytocin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 7/27 | 9/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxytocin (N=27) | Placebo (N=27)
Jitteriness/restlessness (Nervous system disorders) | 4 | 5
Anxiety (Nervous system disorders) | 3 | 3
Dry mouth (Nervous system disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes